CLINICAL TRIAL: NCT06204263
Title: The Effect of the Finger Feeding Method Applied by Fathers on the Transition Time to Oral Feeding and Sucking Success in Premature Babies
Brief Title: The Effect of the Finger Feeding Method Premature Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zülbiye demir barbak, lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AtaU-HEM-ZDB-01
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Premature
Keywords: Premature; Finger; Father; Feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Babies in the control group will be given only routine ward care (breast milk or formula via tube without stimulation of the pacifier or mother's finger).
- Experimental Group (Experimental): The baby will be allowed to suck his father's finger for five minutes three times a day before nasogastric feeding.
  Interventions: Other: finger feeding

INTERVENTIONS:
Other: finger feeding — The fathers of premature babies in intensive care will be interviewed and an educational booklet will be prepared about finger feeding, cleaning, hygiene, hand washing, the importance of sucking, and the rules to be followed to prevent infection in the newborn, and how to apply it will be explained by the researcher. Babies will be breastfed three times a day for seven days.
  Arms: Experimental Group

SUMMARY:
This study aimed to determine the effect of the finger feeding method applied by fathers on the transition time to oral feeding and sucking success in premature babies.

DETAILED DESCRIPTION:
Premature babies followed in the Neonatal Intensive Care Unit will be randomly divided into two groups: control group and finger-feeding group. Babies in the experimental group will be breastfed by their father three times a day. Before nasogastric feeding, the baby will be allowed to suck his finger by putting his finger in his mouth for five minutes three times a day. This procedure will be applied three times a day (morning, noon and evening) for a full 7 days. Babies in the control group will be given only routine ward care (breast milk or formula via tube without stimulation of the pacifier or mother's finger). Preterm Baby Monitoring Form and LATCH Breastfeeding Diagnostic Measurement Tool will be used to determine the transition time to oral feeding and breastfeeding success.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies at 29-31 weeks
* Birth weight of 1300 g or more
* Those whose 1st and 5th minute Apgar scores are over 6
* Those whose vital signs and health status are stable
* In babies who have received mechanical ventilation and continuous positive air pressure support, those who have passed 48 hours after stability has been achieved
* No facial or oral anomalies
* Premature babies without swallowing difficulties
* Those fed via nasogastric tube
* Fathers who can read, write and speak Turkish
* Fathers of preterm babies who agreed to participate in the research.

Exclusion Criteria:

* Those whose vital and health conditions are unstable
* Those whose father has a skin condition or those who developed it later
* Any upper respiratory tract infection in the father
* Premature babies without swallowing difficulties
* Fathers who cannot read, write or speak Turkish
* Fathers with preterm babies who do not consent to this study will not be included in the scope of the research.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Patient Identification Form | Baseline
  This form contains information such as the age of the mother and father, the baby's weight, time to independent oral feeding, discharge weight, length of hospital stay, fetal age at birth, Apgar score, gender of the baby, etc.

SECONDARY OUTCOMES:
Preterm Baby Monitoring Form | Baseline
  During the study process, it will be used to record the preterm baby's "first finger feeding, transition to oral feeding, first latch on the mother's breast, transition to full mother's breast, discharge dates and body weight at these stages, as well as the finger feeding chart" information.

OTHER OUTCOMES:
LATCH Breastfeeding Diagnostic Measurement Tool | Baseline
  It was developed in Oregon by Jensen and Wallace in 1993. LATCH Breastfeeding Diagnosis Form consists of five evaluation criteria: L(Latch on breast), A(Audible swallowing), T(Type of nipple), C(Comfort breast /nipple) and H(Hold / Help) Each item is evaluated between 0-2 points. The lowest score from the scale is 0 and the highest score is 10. High scores indicate the baby's sucking success.

CONTACTS AND LOCATIONS:
Overall Officials: HASAN KAHVECİ, Study Chair — zulbiye.demir@atauni.edu.tr
Locations (1):
- Zülbiye DEMİR BARBAK, Erzurum, Center, Turkey (Türkiye)

REFERENCES:
- [Result] Buldur E, Yalcin Baltaci N, Terek D, Yalaz M, Altun Koroglu O, Akisu M, Kultursay N. Comparison of the Finger Feeding Method Versus Syringe Feeding Method in Supporting Sucking Skills of Preterm Babies. Breastfeed Med. 2020 Nov;15(11):703-708. doi: 10.1089/bfm.2020.0043. Epub 2020 Sep 11. PMID 32915053
- See also: Randomized controlled study — https://pubmed.ncbi.nlm.nih.gov/32915053/